CLINICAL TRIAL: NCT07341841
Title: Assessing Obesity Related Risk Factors in Burke, Columbia, Richmond (BCR) Adult Population: A Genetic and Behavioral Study
Brief Title: Assessing Obesity Related Risk Factors in Adult Population: A Genetic and Behavioral Study
Acronym: ORF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SPH
Record Dates: First submitted 2025-06-13; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Obesity Prevention
Keywords: MC4R, gene variant. obesity, diet
MeSH Terms: interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (Other): Diet and exercise baseline
  Interventions: Behavioral: Diet and exercise; Behavioral: Lifestyle Intervention; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Diet and exercise — Diet intervention: Participants will be randomly divided into a control group (n=50) and a training group (n=50) using the simplest method of assigning participants to different treatment groups: a coin toss. They will be surveyed using the modified DHII questionnaire to assess their caloric intake. The baseline calorie intake will be evaluated during the first visit. Participants will be instructed to reduce their portion sizes by half of what they typically consume. The commitment of participants will be for 8 weeks.
  Exercise intervention: In the first visit, subjects will be familiarized with exercise on a bicycle ergometer to eliminate the novel effects of a new experience. The subjects in the training group will then come to our laboratory to participate in an 8-week exercise program; the control group will not undergo training during this experimental period. The training group will train on a bicycle ergometer for 30 minutes, 3 days a week, for 8 weeks.
Behavioral: Lifestyle Intervention — 8-week personalized diet using a personalized low-calorie diet based on the caloric intake baseline using modified Diet History Questionnaire II (DHQ II)
Behavioral: Exercise — 8-week personalized physical activity- subjects will be doing 30-minute exercise three times a week using a bicycle ergometer

SUMMARY:
This study aims to explore the association between Melanocortin-4 Receptor (MC4R) polymorphisms, eating habits, and social determinants of health in a heterogeneous adult population in Georgia, USA.

DETAILED DESCRIPTION:
The study has three aims.

Aim 1: Genotyping and Participant Stratification To assess the genetic variation of the MC4R gene in the Burke-Columbia-Richmond (BCR) population using Targeted DNA sequencing technology and stratify participants into genotype-based intervention groups (e.g., risk vs. non-risk variants). We anticipate seeing differences in MC4R gene polymorphisms within the BCR residents.

Aim 2: Genotype-Informed Lifestyle Intervention To evaluate the effects of an 8-week personalized dietary and physical activity intervention and association with the frequency distribution of the MC4R variants in the BCR using modified Diet History Questionnaire II (DHQ II) and bicycle ergometer, respectively. In addition, the association between body composition and the subject's age group will be measured using BOD POD instrument. We expect to find associations between food intake and the MC4R variants within the residents of the BCR area. We also expect to see the difference between age groups and the MC4R variant based on body composition.

Primary outcome: change in body composition, primarily body fat percentage Secondary outcomes: changes in dietary patterns, physical activity, and BMI

Aim 3: Socioeconomic and environmental factors To assess whether socio-economic status and environmental inequalities influence diet quality and obesity status of the BCR residents. Data will be collected through a structured questionnaire and secondary sources, such as the U.S. Census Bureau. We expect to find differences in the obesity profiles in the BCR adult population due to socio-economic and environmental inequalities. We hypothesize that the MC4R variants, socio-economic, and environmental inequalities are correlated with eating habits and obesity status within BCR residents.

ELIGIBILITY:
Inclusion Criteria:

Adults 18-70 years old are included in the study.

Target populations are 4 groups:

* Group 1 - overweight (not obese), if BMI is 25.0-29.9 Kg/m2;
* Group 2 - Class 1 (lower-risk) obesity, if BMI is 30.0-34.9 Kg/m2;
* Group 3 - Class 2 (moderate-risk) obesity, if BMI is 35-39.9 Kg/m2 and
* Group 4 - Class 3 (high-risk) obesity, if BMI is equal or greater than 40 Kg/m2.

Males and females will participate in the study.

Exclusion Criteria:

Children younger than 18 years old and adults over 70 are excluded from the study. Non-English speakers and individuals with impaired decision-making capacity to consent are excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Diet and exercise | 8 weeks
  Calorie intake, BMI, % fat, % lean mass.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study